CLINICAL TRIAL: NCT06010433
Title: CERAMENT G Device Registry
Status: Recruiting | Type: Observational
Sponsor: BONESUPPORT AB (Industry)
Responsible Party: Sponsor
Other Study IDs: S050/2018
Record Dates: First submitted 2023-05-25; First posted 2023-08-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Osteomyelitis; Fracture Related Infection; Diabetic Foot Osteomyelitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CERAMENT G — * Primary mode of action is to be a resorbable ceramic bone graft substitute intended to fill gaps and voids in the skeleton system to promote bone healing. CERAMENT ™|G provides a void/gap filler that during the surgical procedure can augment hardware and bone alignments.
  * Secondary mode of action is to prevent colonization of Gentamicin sensitive microorganisms in order to protect bone healing.

SUMMARY:
This is an Observational Device Registry Study of CERAMENT|G in normal use in accordance with the IFU. It will run for a period of three years from enrolment of the first patient into the Study at each Site, before being subject to review. A Device Registry is a form of observational study that concerns the performance of a device in normal use. It is intended to collect data that is reflective of 'real world' device performance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over (on the day of surgery)
* receive CERAMENT|G as a component of their treatment at a participating, contracted centre or healthcare provider, in accordance with the IFU for the implanted product
* In receipt of patient information leaflet and have signed appropriately designed informed consent form.

Exclusion Criteria:

* Any exclusion criteria as per IFU for CERAMENT|G
* Any off-label use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The racial, gender and ethnic characteristics of the individuals approached for participation in this Observational Registry Study shall reflect the demographics of patients that would ordinarily receive CERAMENT|G for the treatment of their condition at the designated investigative centres. No individuals shall be excluded from participation in the Observational Registry Study based on race, nationality, ethnicity, gender, or sexuality
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2028-09-22 (Estimated); Study Completion 2028-09-22 (Estimated)

PRIMARY OUTCOMES:
Primary Outcomes | 12 months
  • Device safety - any unexpected device performance, complaints, adverse events, adverse device effects, SAEs throughout study period.

SECONDARY OUTCOMES:
Secondary Outcome | 12 months
  Bone healing at final follow-up
Secondary Outcome | 6 and 12 months
  Pain and functional assessment at whatever follow-up times are usual for the specific clinical site, for example 6 & 12 months, if normally conducted
Secondary Outcome | 12 months
  (Recurrence of) infection/revision surgery

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - North Park Podiatry, San Diego, California
  - OrthoCarolina, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No